CLINICAL TRIAL: NCT05767164
Title: Correlation Between Parameters and Prognosis of Cervical Single Open-door Surgery: a Multicenter Retrospective Clinical Study
Brief Title: Correlation Between Parameters and Prognosis of Cervical Single Open-door Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Xi'an Honghui Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KY20222157-C-1
Record Dates: First submitted 2023-02-18; First posted 2023-03-14 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Cervical Spinal Stenosis
Keywords: Cervical single open-door surgery; Cervical Spinal Stenosis; Open angle

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Preoperative (No Intervention)
- postoperative (3 months) (Experimental)
  Interventions: Procedure: cervical single open-door surgery
- postoperative (6 months) (Experimental)
  Interventions: Procedure: cervical single open-door surgery
- postoperative (1 year) (Experimental)
  Interventions: Procedure: cervical single open-door surgery

INTERVENTIONS:
Procedure: cervical single open-door surgery — The patients were operated by the cervical single open-door surgery, which were used with the Centerpiece titanium plate to internal fixation.
  Arms: postoperative (1 year); postoperative (3 months); postoperative (6 months)

SUMMARY:
The aim of study was evaluated the relationship between the relevant evaluation indexes of cervical spine open-door surgery, prognosis and complication rate, and provided theoretical basis for personalized surgical program through multi-center retrospective clinical study

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of the patients were typical. MRI showed single or multiple central herniation of C3-C7 intervertebral discs or spinal stenosis at corresponding levels, which confirmed cervical myeloid cervical spondylosis or cervical spinal stenosis.
* Conservative treatment for more than 3 months before surgery was ineffective.
* The patients underwent cervical single open-door surgery.
* Informed consent was obtained from the patient and his family, informed consent was signed, and a complete follow-up was completed after surgery

Exclusion Criteria:

* Cervical spondylotic radiculopathy.
* Cervical kyphosis or instability.
* Cervical spondylosis caused by trauma, tumor, tuberculosis and metabolic diseases.
* Revision surgery or combined anterior-posterior surgery is required.
* The patients had severe neurological diseases affecting the evaluation of postoperative results.
* Psychopath.
* MRI or CT for contraindications.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
lamina open angle | 3 months after surgery
  The Angle of opening of the cervical unilateral lamina while cervical single open-door surgery
JOA score change | pre-operation,3 months after surgery, 1 year after surgery
  Japanese Orthopedic Association (JOA) score is used to assess the function of spinal cord which is in the form of questionnaires. Postoperative improvement rate = ((postoperative score - preoperative score)/ (17- preoperative score)) X100%. Improvement rate can also correspond to the commonly used efficacy criteria: cure when the improvement rate is 100%, effective when the improvement rate is greater than 60%, effective when 25-60%, and ineffective when less than 25%.
NDI score change | pre-operation,3 months after surgery, 1 year after surgery
  Neck Disability Index (NDI) score is used to assess the disorder of spinal cord which is in the form of questionnaires. Postoperative improvement rate = (total score)/ (numbers of programme X5) X100%. Improvement rate can also correspond to the commonly used efficacy criteria: the improvement rate when 60%-80% means extremely severe dysfunction, when 40%-60% means severe dysfunction, when 20-40% means moderate dysfunction, and when less than 20% means mild dysfunction.
VAS score change | pre-operation,3 months after surgery
  A Visual Analogue Scale (VAS) is used to measure the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. Using a ruler, the score is determined by measuring the distance (mm) on the 10cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Maximum spinal cord compression change | pre-operation,3 months after surgery, 1 year after surgery
  This index was measured by MRI, which was the ratio of the diameter of the cervical pulp at the most compressed segment to the mean diameter of the cervical pulp at the upper and lower segments without compression
Compression ratio change | pre-operation,3 months after surgery, 1 year after surgery
  This index was measured by MRI, which means the minimum sagittal diameter of the cervical pulp in the most compressed segment divided by maximum transverse diameter
transverse area change | pre-operation,3 months after surgery, 1 year after surgery
  This index was measured by MRI, which means the cross-sectional area of the cervical pulp at the highest level of compression.
Sagittal Canal Diameter change | pre-operation,3 months after surgery, 1 year after surgery
  This index was measured by CT, which was sagittal diameter of the spinal canal at the most compressed level.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shannxi Province, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hirabayashi K, Miyakawa J, Satomi K, Maruyama T, Wakano K. Operative results and postoperative progression of ossification among patients with ossification of cervical posterior longitudinal ligament. Spine (Phila Pa 1976). 1981 Jul-Aug;6(4):354-64. doi: 10.1097/00007632-198107000-00005. PMID 6792717
- [Background] Karpova A, Arun R, Davis AM, Kulkarni AV, Massicotte EM, Mikulis DJ, Lubina ZI, Fehlings MG. Predictors of surgical outcome in cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2013 Mar 1;38(5):392-400. doi: 10.1097/BRS.0b013e3182715bc3. PMID 23448898
- [Background] Nouri A, Tetreault L, Zamorano JJ, Dalzell K, Davis AM, Mikulis D, Yee A, Fehlings MG. Role of magnetic resonance imaging in predicting surgical outcome in patients with cervical spondylotic myelopathy. Spine (Phila Pa 1976). 2015 Feb 1;40(3):171-8. doi: 10.1097/BRS.0000000000000678. PMID 25668335
- [Background] Torg JS, Pavlov H, Genuario SE, Sennett B, Wisneski RJ, Robie BH, Jahre C. Neurapraxia of the cervical spinal cord with transient quadriplegia. J Bone Joint Surg Am. 1986 Dec;68(9):1354-70. PMID 3782207
- [Background] Yeh KT, Lee RP, Chen IH, Yu TC, Liu KL, Peng CH, Wang JH, Wu WT. Laminoplasty instead of laminectomy as a decompression method in posterior instrumented fusion for degenerative cervical kyphosis with stenosis. J Orthop Surg Res. 2015 Sep 4;10:138. doi: 10.1186/s13018-015-0280-y. PMID 26338009
- [Background] Pavlov H, Torg JS, Robie B, Jahre C. Cervical spinal stenosis: determination with vertebral body ratio method. Radiology. 1987 Sep;164(3):771-5. doi: 10.1148/radiology.164.3.3615879.
- [Background] Blackley HR, Plank LD, Robertson PA. Determining the sagittal dimensions of the canal of the cervical spine. The reliability of ratios of anatomical measurements. J Bone Joint Surg Br. 1999 Jan;81(1):110-2. doi: 10.1302/0301-620x.81b1.9001. PMID 10068016
- [Background] Prasad SS, O'Malley M, Caplan M, Shackleford IM, Pydisetty RK. MRI measurements of the cervical spine and their correlation to Pavlov's ratio. Spine (Phila Pa 1976). 2003 Jun 15;28(12):1263-8. doi: 10.1097/01.BRS.0000065570.20888.AA. PMID 12811269